CLINICAL TRIAL: NCT02534818
Title: Conventional Fluorescein Sodium Dosage o.1ml/kg Compared With a Lower Fluorescein Sodium Dosage o.02ml/kg for the Detection of Gastric Intestinal Metaplasia in a High Risk Population: a Randomized Controlled Trial
Brief Title: Different Fluorescein Sodium Dosage for the Detection of Gastric Intestinal Metaplasia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015SDU-QILU-G09
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): lower fluorescein sodium dosage 0.02ml/kg for gastric intestinal metapalsia
  Interventions: Drug: lower fluorescein sodium dosage 0.02ml/kg
- Group 2 (Active Comparator): conventional fluorescein sodium dosage 0.1ml/kg for gastric intestinal metapalsia
  Interventions: Drug: conventional fluorescein sodium dosage 0.1ml/kg

INTERVENTIONS:
Drug: lower fluorescein sodium dosage 0.02ml/kg — fluorescein Sodium Dose of 0.02ml/kg on gastric intestinal metapalsia
  Arms: Group 1
Drug: conventional fluorescein sodium dosage 0.1ml/kg — fluorescein Sodium Dose of 0.1ml/kg on gastric intestinal metapalsia
  Arms: Group 2

SUMMARY:
The purpose of this study is to assess whether lower fluorescein sodium dosage can perceive the same detection rate per patient and per lesion for the detection of gastric intestinal metaplasia.

DETAILED DESCRIPTION:
Gastric intestinal metaplasia is regarded as an important premalignant lesion for intestinal type gastric cancer. Currently, the histological assessment of gastric intestinal metaplasia still relies on the biopsies took from five sites that the updated Sydney System recommended.

This study aims to compare the diagnostic yield of gastric intestinal metaplasia from two different fluorescein sodium dosage and assess whether lower fluorescein sodium dosage can perceive the same detection rate per patient and per lesion for the detection of gastric intestinal metaplasia.

ELIGIBILITY:
Inclusion Criteria:

* patients with dyspeptic symptoms and aged 40 years or older
* or patients with Helicobacter pylori infection, or histologically verified gastric intestinal metaplasia or atrophic gastritis
* or patients with family history of gastric cancer

Exclusion Criteria:

* presence of gastrectomy, acute gastrointestinal bleeding, or known gastric neoplasia
* presence of conditions unsuitable for endoscopy procedure including coagulopathy, impaired cardiopulmonary function , pregnancy or breastfeeding
* inability to provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Difference of the detection rate of gastric intestinal metaplasia between two fluosecein sodium dosage in a per-pateint analysis | six months
Difference of the detection rate of gastric intestinal metaplasia between two dosage fluosecein sodium in a per-biopsy analysis | six months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD, Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China